CLINICAL TRIAL: NCT00555971
Title: A Placebo Controlled, Double-Blind Investigation of the Therapeutic Utility of Xolair (Omalizumab) for Attenuating Aspirin Induced Bronchospasm in Patients With Aspirin Exacerbated Respiratory Disease (AERD) Undergoing Aspirin Desentization
Brief Title: Therapeutic Utility of Xolair in Patients Undergoing Aspirin Desensitization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David Lang (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David Lang, Chairman, Allergy and Immunology, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 05-066; Q3637s (Other Grant/Funding Number: Genentech)
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Aspirin Sensitivity
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Group (Placebo Comparator): Subjects randomized to placebo
  Interventions: Drug: placebo
- Omalizumab Group (Active Comparator): Subjects randomized to omalizumab
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Subjects randomized to Omalizumab prior to aspirin desensitization
  Other Names: Xolair
  Arms: Omalizumab Group
Drug: placebo — Subjects randomized to Placebo prior to aspirin desensitization
  Arms: Placebo Group

SUMMARY:
This is a 24 week double-blind study in which subjects will be randomized 2:1 to receive Xolair (Omalizumab) or placebo. 14 subjects will receive Xolair and 7 will receive placebo. Xolair injections will occur every 2-4 weeks. Aspirin desensitization will occur several weeks later. One month after desensitization, the final visit will occur in the GCRC.

We hypothesize that administration of Xolair, a monoclonal anti-IgE antibody, prior to the aspirin desensitization will reduce severity of aspirin-induced reaction.

DETAILED DESCRIPTION:
This is a 24 week double-blind study consisting of up to 11 office visits for people 18 years of age with aspirin exacerbated respiratory disease (AERD). 21 subjects will participate and will be randomized 2:1 to receive Xolair (Omalizumab) or placebo. 14 subjects will receive Xolair and 7 will receive placebo. Xolair is a FDA approved medication for the treatment of moderate to severe allergic asthma. Injections will occur every 2-4 weeks, for 16 weeks. The dosage will be based upon IgE and body weight. Aspirin desensitization will occur 1-3 weeks later. One month after desensitization, the final visit will occur in the GCRC.

Properly selected patients with aspirin exacerbated respiratory disease (AERD) experience benefit in the course of their disease with aspirin desensitization treatment; however, AERD patients are at risk for potentially serious asthmatic reaction when undergoing aspirin desensitization. For this reason, this procedure is currently performed in a monitored setting. We hypothesize that administration of Xolair, a monoclonal anti-IgE antibody, prior to the aspirin desensitization will reduce severity of aspirin-induced respiratory reaction, and that ultimately, use of Xolair will permit this procedure to be performed safely in outpatient settings. This protocol also entails obtaining blood and urine samples to assess the influence of Xolair, compared with placebo. As aspirin induced reaction occurs via heightened release of leukotrienes combined with greater end organ responsiveness to these mediators, we also will be quantifying the impact of prior administration of Xolair, compared with placebo, on the elevation of urinary LTE4 in association with aspirin challenge and with aspirin provoked reaction.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Fulfill diagnostic criteria for AERD (described below), and be a candidate for aspirin desensitization chronic asthma - frequently moderate-severe or severe patients will have history compatible with variable airflow obstruction. chronic rhinosinusitis - usually requiring previous sinus surgery procedure(s). sinusitis will have been confirmed by imaging studies presently and/or in the past.

history of adverse reaction to aspirin and/or aspirin-like drugs (e.g., ibuprofen, naproxen, etc.) compatible with AERD.

• Candidate for Xolair [Omalizumab] Moderate-severe persistent asthma IgE = 30-700 IU/ml IgE mediated (allergic) potential to inhalant allergen(s) by cutaneous or in vitro testing.

Exclusion Criteria:

* Women of childbearing potential not using appropriate contraception method(s)
* Women currently breastfeeding
* Women who desire to become pregnant during the time of participation in this study
* Men who desire to get someone pregnant during participation in this study
* Known sensitivity to Xolair [Omalizumab].
* IgE level < 30 IU/ml, or > 700 IU/ml.
* No evidence of atopy by immediate hypersensitivity skin testing
* Use of any other investigational agent in the last 30 days
* Age < 18 years.
* Current tobacco habituation.
* Presence of emphysema
* Ethanolism or drug abuse within last 12 months.
* Presence of significant medical condition including malignancy, neurologic, kidney, gastrointestinal, liver or cardiovascular disease
* extensive travel commitments during the study that would interfere with study measurements or clinic visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Lang, M.D., Principal Investigator — The Cleveland Clinic, Department of Allergy and Immunology
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lang DM, Aronica MA, Maierson ES, Wang XF, Vasas DC, Hazen SL. Omalizumab can inhibit respiratory reaction during aspirin desensitization. Ann Allergy Asthma Immunol. 2018 Jul;121(1):98-104. doi: 10.1016/j.anai.2018.05.007. Epub 2018 May 16. PMID 29777744

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients seen for evaluation and management for suspected AERD
Pre-assignment Details: 16 subjects signed consent but only 13 were randomized 2 were screen fails and 1 lost to follow up
Groups:
- Placebo: Subjects with aspirin exacerbated respiratory disease enrolled and randomized to either omalizumab or placebo (2:1) in a blinded fashion, administered for 16 weeks. The study is double-blind.
  placebo: aspirin desensitization will be carried out for all subjects with aspirin exacerbated respiratory disease who participate in the study, with subjects randomized 2:1 to receive either omalizumab or placebo, which will allow us to evaluate the study hypothesis
- Omalizumab: Subjects with aspirin exacerbated respiratory disease enrolled and randomized to either omalizumab or placebo (2:1) in a blinded fashion, administered for 16 weeks. The study is double-blind.
  Omalizumab: aspirin desensitization will be carried out for all subjects with aspirin exacerbated respiratory disease who participate in the study, with subjects randomized 2:1 to receive either omalizumab or placebo, which will allow us to evaluate the study hypothesis
Period: Overall Study
Arm/Group | Placebo | Omalizumab
Started | 5 | 8
Completed | 4 | 7
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omalizumab | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (7.2) | 45.7 (11.9) | 44.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
FEV1 Percent predicted [Mean (Standard Deviation); unit: Percent predicted] — Lung function measurement
  Percent predicted | 90.0 (18.5) | 92.6 (14.4) | 91.6 (16.8)
IgE IU/ml [Mean (Standard Deviation); unit: IU/ml] | 64.6 (36.6) | 120.5 (76.7) | 100.3 (73.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Respiratory Reaction During Aspirin Desensitization
Description: Lack of Respiratory reaction during aspirin desensitization, including Spirometry (FEV1) testing, to assess the efficacy of Xolair on attenuating aspirin induced bronchospasm in patients with AERD.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 4 | 7
Participants | 0 | 5
Statistical Analysis 1: Comparison: Placebo vs Omalizumab; Test type: Equivalence — This was a statistical analysis to address the null hypothesis that there was no difference between treatment and placebo groups; p = 0.036, Fisher Exact

2. Secondary Outcome: Measurements of Urinary LTE4 in Association With Respiratory Reaction During Aspirin Desensitization
Description: Measurements of urinary LTE4 in association with aspirin desensitization, comparing subjects randomized to placebo with subjects randomized to omalizumab, with study drug administered for 16 weeks. Measurements were compared for respiratory reaction in placebo subjects who exhibited either upper or lower airway reaction and after 100 mg aspirin challenge dose in omalizumab subjects who were non-reactors. For this analysis, the two omalizumab subjects who had respiratory reaction were not included.
Time Frame: Approximately 24 weeks
Measure: Mean (Standard Error); unit: pg/mg creatinine units
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 4 | 5
pg/mg creatinine units | 17489 (7102) | 1852 (280)

ADVERSE EVENTS:
Time Frame: Entire study until last randomized subject completed participation, approximately 24 weeks
Arm/Group | Placebo | Omalizumab
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 1/4 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Omalizumab (N=7)
Aspirin intolerance (Gastrointestinal disorders) | 1 (1) | 0 (0) — A subject in Phase D developed gastrointestinal intolerance, was instructed to suspend aspirin, and did not complete study participation.

LIMITATIONS AND CAVEATS:
Findings cannot be generalized to patients with aspirin exacerbated respiratory disease receiving omalizumab for less than 16 weeks, or to those who do not fulfill label criteria for omalizumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2013-01-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT00555971/Prot_000.pdf